CLINICAL TRIAL: NCT06867601
Title: Healthcare Professionals in German Psychiatric-psychosomatic Clinical Practice: Theory Guided Evaluation of Work-related Challenges.
Brief Title: Work-related Challenges in Psychiatric-psychosomatic Clinics
Acronym: HIPP
Status: Recruiting | Type: Observational
Sponsor: Jacobs University Bremen gGmbH (Other)
Responsible Party: Sponsor
Other Study IDs: HIPP_27112024
Record Dates: First submitted 2025-02-26; First posted 2025-03-10 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Work Engagement; Burnout; Job Satisfaction; Turnoverintention; Service Quality
Keywords: Health Care Providers; Patient Safety; Occupational well-being
MeSH Terms: conditions — Burnout, Psychological

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Nurses
- Psychologists
- Doctors (Psychiatrists)

SUMMARY:
The aim of this project is to evaluate the work-related challenges faced by healthcare professionals (nurses, psychologists, and doctors) in German psychiatric-psychosomatic clinics. By applying the Job Demands-Resources (JD-R) model, this study investigates how job demands and resources influence job satisfaction, turnover intention, and subjective service quality. Special focus is given to the roles of burnout, engagement, and psychological safety as mediators and moderators in these relationships. Through a cross-sectional online survey targeting 600 healthcare professionals, this study aims to identify key factors affecting well-being and performance in mental health settings. The findings will contribute to the development of interventions to improve the working conditions and service quality in psychiatric-psychosomatic care.

DETAILED DESCRIPTION:
This study uses an online questionnaire to collect data from healthcare professionals (nurses, psychologists, and doctors) working in psychiatric-psychosomatic clinics in Germany. The survey aims to assess their experiences and perceptions regarding work-related challenges, job demands, and resources, as well as their impact on job satisfaction, turnover intention, and subjective service quality. The study applies the Job Demands-Resources (JD-R) model to explore the relationships between these factors, with a particular focus on the mediating roles of burnout and engagement and the moderating role of psychological safety.

The survey will be conducted at a single time point, targeting 600 healthcare professionals (200 nurses, 200 psychologists, and 200 doctors) across various psychiatric-psychosomatic clinics in Germany. Data will be collected using standardized scales to ensure reliability and validity. Participants will be recruited via email invitations sent to clinics, with the survey distributed through the SoSci Survey platform. Participation is voluntary, and all data will be anonymized and handled in compliance with ethical and data protection regulations.

Main Research Questions are:

I. How do the surveyed resources and demands of healthcare professionals impact job satisfaction, turnover intention and subjective service quality? II. What roles do burnout, engagement, and psychological safety play as mediators and moderators in these relationships? III. What are the key challenges and resources identified by healthcare professionals in their daily work within psychiatric-psychosomatic settings?

ELIGIBILITY:
Inclusion Criteria:

* Healthcare professionals (nurses, psychologists, or doctors) working in psychiatric-psychosomatic clinics in Germany
* Age 18 years or older
* Sufficient German language proficiency to complete the questionnaire
* Willingness to provide informed consent

Exclusion Criteria:

* Individuals not working as nurses, psychologists, or doctors in psychiatric-psychosomatic clinics
* Age under 18 years
* Insufficient German language proficiency to complete the questionnaire
* Massively limited cognitive abilities

Ages: 18 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Healthcare professionals (nurses, psychologists, and doctors) working in German psychiatric-psychosomatic clinics
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2025-03-10 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Job Satisfaction | Baseline
  The 'Arbeitszufriedenheit Skala' (Job Satisfaction Scale) from the Copenhagen Psychosocial Questionnaire (COPSOQ) by Nübling et al. (2010) assesses job satisfaction among healthcare professionals in psychiatric-psychosomatic clinics. This scale captures various dimensions of job satisfaction, including satisfaction with career prospects, colleagues, physical working conditions, management, utilization of skills, salary, and overall job satisfaction. Responses are measured on a 5-point Likert scale, ranging from 1 (Very satisfied) to 5 (Very dissatisfied). Higher scores indicate lower job satisfaction, while lower scores reflect higher job satisfaction.
Emotional Exhaustion | Baseline
  The 'Emotionale Erschöpfung Skala' (Emotional Exhaustion Scale) from the Copenhagen Psychosocial Questionnaire (COPSOQ) by Nübling et al. (2010) assesses emotional exhaustion among healthcare professionals in psychiatric-psychosomatic clinics. This scale captures participants' experiences of exhaustion and feelings of being emotionally drained due to work. Responses are measured on a 5-point frequency scale, ranging from 1 (Always) to 5 (Never/Almost never). Lower scores indicate greater emotional exhaustion, while higher scores reflect lower levels of exhaustion.
Engagement | Baseline
  The 'Engagement Skala' from the Copenhagen Psychosocial Questionnaire (COPSOQ) by Nübling et al. (2010) assesses work engagement among healthcare professionals in psychiatric-psychosomatic clinics. They collect data on participants' levels of energy, enthusiasm, and absorption in their work. Responses are measured on a 5-point frequency scale ranging from 1 (Always) to 5 (Never/Almost never). Lower scores indicate grater engagement, while higher scores reflect lower levels of engagement.

SECONDARY OUTCOMES:
Turnover Intention | in the last 12 Months
  The 'Gedanke an Beruf-/Stellenwechsel Skala' (Turnover Intention Scale) from the Copenhagen Psychosocial Questionnaire (COPSOQ) by Nübling et al. (2010) assesses turnover intention among healthcare professionals in psychiatric-psychosomatic clinics. They collect data on participants' thoughts about leaving their profession or their current job over the past 12 months. Responses are measured on a 5-point frequency scale ranging from 1 (Never) to 5 (Every day). Lower scores indicate a lower desire to leave the job, while higher scores reflect greater desire to leave.
Subjective Service Quality | Baseline
  The 'Service Quality Scale' by Rafferty et al. (2001) assesses subjective service quality among healthcare professionals in psychiatric-psychosomatic clinics. They collect data on participants' perceptions of the quality of care provided on their unit, including reliability, consistency, and alignment with expectations. Responses are measured on a 5-point Likert scale ranging from 1 (Strongly disagree) to 5 (Strongly agree). Lower scores indicate a subjective lower service quality, while higher scores reflect higher subjective service quality.

CONTACTS AND LOCATIONS:
Overall Officials: Sonia Lippke, Prof. Dr., Study Director — Constructor University Bremen gGmbH & Bremen International Graduate School of Social Sciences, Germany
Locations (2):
- Germany (2):
  - Constructor University Bremen and online, Bremen, City state Bremen
  - Constructor University, Bremen, City state Bremen